CLINICAL TRIAL: NCT05802472
Title: Effect of Polyphenolic Extract of Vachellia Farnesiana on Glycemic Response and Safety in Healthy Volunteers.
Brief Title: Effect of an Polyphenolic Beverage in Healthy Volunteers
Acronym: PB
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, Claudia Delgadillo Puga, Dr, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 3910
Record Dates: First submitted 2023-03-15; First posted 2023-04-06 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-01

CONDITIONS: Healthy; Safety Issues
Keywords: Randomized single-blind clinical trial; Vachellia farnesiana; polyphenolic beverage; Phase I

STUDY DESIGN:
Intervention Model Description: Single-blind, placebo-controlled, randomized clinical trial.
Who Masked: Participant
Masking Description: Block randomization. This procedure aims to ensure a periodic balance in the number of subjects assigned to each intervention group (53). The size of each block will be six individuals, and the number of blocks will be 10; the permutation of the groups was defined as Control (C) and Experimental (E). It is important to note that the blocks and permutations were randomly assigned.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Placebo Comparator): Thirty subjects were randomly assigned (Visit 1), and weight and height will be evaluated, as body composition, and blood sampling to assess glucose, liver, and kidney function. During Visit 2, and before the administration of a single water as placebo, glucose in the blood will be quantified (basal; with 12 hours of fasting); later, administer a load of 75 g of oral sucrose and after 30 minutes, the blood sample will begin at different intervals: 20, 40, 60, 90 and 120 minutes. The participant solves the food consumption frequency questionnaires during this procedure. A second blood sample will be taken 48 hours later (Visit 3). Finally, a urine sample will be taken to rule out acute kidney damage through the sensitive kidney damage biomarker (KIM-1). In addition, the participant will be interviewed to answer the adverse effects questionnaire.
  Interventions: Other: Polyphenolic beverage from extract of Vachellia farnesiana
- Experimental beverage group (Experimental): Thirty subjects were randomly assigned (Visit 1), and weight and height will be evaluated, as body composition and blood sampling to assess glucose, liver, and kidney function. During Visit 2, and before the administration (1.2 mg/kg of weight) of a single infusion of the polyphenolic extract, glucose in the blood will be quantified (basal; with 12 hours of fasting); later, administer a load of 75 g of oral sucrose and after 30 minutes, the blood sample will begin at different intervals: 20, 40, 60, 90 and 120 minutes. The participant solves the food consumption frequency questionnaires during this procedure. A second blood sample will be taken 48 hours later (Visit 3). Finally, a urine sample will be taken to rule out acute kidney damage through the sensitive kidney damage biomarker (KIM-1). In addition, the participant will be interviewed to answer the adverse effects questionnaire.
  Interventions: Other: Polyphenolic beverage from extract of Vachellia farnesiana

INTERVENTIONS:
Other: Polyphenolic beverage from extract of Vachellia farnesiana — During Visit 2. A single infusion of the polyphenolic extract was administered orally. The dose (1.2 mg/kg body weight) of lyophilized extract, which was diluted in water, was calculated considering each participant's weight.

SUMMARY:
Currently, there are different strategies to prevent the effect of beverages and foods on blood glucose levels after ingestion. In this sense, polyphenols are a promising field; these compounds are secondary metabolites produced by plants, vegetables, and fruits; of these compounds, gallic acid, quercetin, and kaempferol stand out for their antihyperglycemic characteristics through a) complex formation, b) enzymatic inhibition, c) affecting transport and, d) stimulation of the secretion of intestinal satiety hormones. Vachellia farnesiana (VF) is a shrub distributed in arid, semi-arid, and tropical regions of Mexico and the world. The polyphenols of the fruits of VF in pre-clinical studies by this research group have shown important antioxidant activity and antihyperglycemic effects. The present proposal aims to evaluate the effect of the polyphenolic extract of Vachellia farnesiana on glycemic response and to monitor liver and renal function tests as a safety control in healthy volunteers through developing a Phase I clinical study.

DETAILED DESCRIPTION:
The increased consumption of high carbohydrate, processed, and non-fiber foods increases the risk of obesity and consequently the development of type 2 Diabetes Mellitus (DM2); therefore, one of the approaches in the prevention and treatment of these diseases has been focused on the management and reduction of the rate of absorption and metabolism of carbohydrates. DM2 is the result of chronic insulin resistance and loss of pancreatic ß-cell mass and function, which may be caused by glucotoxicity and lipotoxicity leading to apoptosis and dysfunction of these cells; the search for alternative therapies has focused research on secondary compounds from plant metabolism, particularly polyphenols (flavonoids), which have shown positive effects on postprandial blood glucose reduction (2). Polyphenols, defined as secondary metabolites produced by plants, can be found in flowers, vegetables, and fruits; they are generated as a defense mechanism against stress, cold, and UV radiation, among other factors. Polyphenols are classified into two large groups: 1) flavonoids and 2) non-flavonoids. An aromatic ring with a hydroxyl group characterizes the structure of polyphenols.

The consumption of polyphenolics around the world is highly variable; it has been reported that in France, the average consumption is between 283 and 1000 mg/day; in Spain, between 500 and 1000 mg/day; in Italy, it is close to 700 mg/day, and in South Korea an average of 320 mg/day, among others. The variety of dietary patterns worldwide will depend on the total amount of polyphenols consumed daily. The consumption of anthocyanins has been associated with preventing and managing DM2 by protecting against pancreatic beta-cell oxidation, decreasing carbohydrate digestion enzymes, and inhibiting advanced glycation products. Over time, polyphenols have been investigated in several experimental models and clinical trials, contributing to the knowledge of their application as potential preventive agents and in the treatment of chronic non-communicable diseases.

One of the essential compounds in this evidence is gallic acid; this polyphenol is found in vegetables, fruits, tea, and red wine; important biological activities have been reported in murine models in metabolic diseases such as DM2, in addition to the regulation of the peroxisome proliferation receptor (PPAR) in liver, muscle and adipose tissue; impacting on the reduction of serum glucose. Furthermore, in vitro studies have documented a crucial inhibitory activity of glycogen phosphorylase enzymes, which participates in the regulation of glycogen metabolism; a strategy that could be used as an antihyperglycemic agent, and another method could focus on the reduction of the alpha-glucosidase enzyme, which participates by reducing carbohydrate absorption at the intestinal level.

The study of another flavonoid present in tomatoes, tubers, oranges, apples, green and black tea, potatoes, and in plants such as Vachellia farnesiana has been quercetin; this component is mainly absorbed in the intestine with low intensity in the portal vein. In subjects with DM2, this compound showed a decrease in serum glucose peaks after administering a single dose of 200 mg of quercetin, a phenomenon that extended during the three hours of follow-up of glucose concentration compared to the placebo group. A meta-analysis reported that oral administration of quercetin >500 mg/day for eight weeks decreased fasting plasma glucose concentration in patients with metabolic syndrome. In another trial, quercetin was administered for eight weeks at 250 mg/day in patients with DM2, significantly decreasing LDL levels and increasing total antioxidant capacity. However, it showed no change in plasma glucose compared to a placebo group, suggesting that the dose was insufficient. Other compounds identified with antihyperglycemic effects are caffeic, gallic, ferulic, and vanillic acids, flavones (rutin), and flavanones (naringenin).

Glucose uptake in peripheral tissues can be affected by the presence of polyphenol compounds through different effects such as: 1) inhibition of monoglyceride digestive enzymes (alpha-amylase and alpha-glucosidase), these digestive enzymes will decrease glucose uptake and 2) reduction of glucose uptake through inhibition of sodium-dependent glucose transporters 1 (SGLT1) and 2 (SGLT2) located in the proximal tubules of the kidney, 3) in addition to stimulation of insulin secretion and protection of beta-pancreatic cells 4) and finally through inhibition of SGLT2 transporters located not only in the renal tubules; but also in other tissues.

Evaluating the safety of polyphenol consumption is essential, so the findings or antecedents available both in vitro and in vivo are considered. Polyphenols have different physiological functions; it is necessary to evaluate the safety of administration; evidence of acute toxicity and clinical toxicity is presented by considering biochemical tests such as liver function and renal function tests. Some weight loss supplements given as plant extracts have been related to acute hepatic injury. Its main component is hydroxy citric acid; some cases report an elevation of transaminases and total bilirubin.

The results that have been generated in pre-clinic studies by the INCMNSZ research team facilitated the calculation to determine an initial dose to be evaluated in the following clinical phase in humans; it is necessary to perform the analysis transferred from mouse to humans calculated by the formula of "transferred dose based on body surface area (BSA)," considering both the weight and the height of an average individual with 60 kg of weight. An initial dose of 1.2 mg/kg of VF extract was calculated for testing; Reagan-Shaw and coworkers described the calculation methodology extensively. However, the average estimated dose should be adjusted using the individual values of weight and height of each participant to determine the surface area of the BSA body.

This phase I clinical study is based on the preclinical tests performed by the INCMNSZ team to determine the No-Observed-Adverse-Effect-Levels (NOAELs), where the dose transferred from mouse to Human; was based on the recommendations of the Food and Drug Administration (FDA) in 2005, where the mouse-human conversion equations are used; it is also recommended to use the value of the body surface area to calculate the human equivalent dose (HED, Human Equivalent Dose) proposed by Nair and Jacob in 2016. In this sense, as part of the research development of dietary alternatives to mitigate the metabolic alterations of obesity from the fruits of VF in male C57BL6 mice, we have established that a dose of 10 mg/kg mouse weight can be transferred, for preclinical studies, as this proposal.

Maintaining glucose homeostasis is of the most physiological importance and is governed by strict hormonal control. The malfunctioning of these hormones can trigger different alterations, such as energy homeostasis disorders that include obesity, hyperglycemia, and glucose intolerance that trigger diseases such as DM2. The influence of polyphenols on the bioavailability of macronutrients plays an important role. It has been reported that they can form complexes with polysaccharides affecting the insulinemic and glycemic response and increasing the excretion of nitrogen and fat in fecal material; they can also suppress the release of glucose from the liver and improve glucose uptake in peripheral tissues. Flavonoids present in vegetables or plants are found in the form of glycosides. These glycosides are hydrolyzed by an enzyme of the ß-glucosidase group (lactase phlorizin hydrolase) located at the brush border of the small intestine, leaving the flavonoid glycoside free; these can subsequently go through the cell membrane by passive diffusion or can be absorbed intact through the sodium-dependent glucose transporters SGLT1. Metabolism of polyphenols begins in the intestinal lumen; they are deconjugated by the lactase phloridzin hydrolase, then the flavonoid is conjugated by uridine diphosphate glucuronyl transferases, and the conjugates exported back into the lumen or blood by various transporters. In addition, metabolites can be transported into hepatocytes via various uptake transporters and then returned to the circulatory system. Alternatively, they can be deconjugated intracellularly by enzymes such as β-glucuronidase and excreted by the kidney. This involves transporters' uptake into proximal tubular cells and excretion in the urine. Still, these transformations depend on the conditions of each individual; some are increased in inflammatory processes. It is essential to mention that although preclinical studies of FV do not show any adverse effects, evaluating its safety in clinical trials for subsequent clinical application is critical. Most clinical studies start without exploring the possible toxic effects of polyphenol consumption. Epigallocatechin compounds have been shown to have a potential prooxidant action which may have implications concerning toxicity and suggest that further research into liver and renal toxicity should be done. There are several recent case reports of hepatotoxicity related to the consumption of high doses of tea-based dietary supplements. In almost all cases (eight out of nine), patients had elevated serum alanine aminotransferase and bilirubin levels. In two of the nine points, periportal and portal inflammation was observed. All cases were resolved after cessation of supplementation. Liver and kidney toxicity have been proposed to be associated with the compound's bioavailability. Recent human studies have shown that fasting increases the bioavailability of some polyphenols, such as epigallocatechin. Although there are no reports of toxicity in volunteers in intervention studies, careful monitoring of liver and kidney function is required until the risk of toxic events associated with tea catechins in humans is established.

Vachellia farnesiana (VF) is a shrub of the Fabaceae family; it is distributed in arid, semi-arid, and tropical regions in Mexico and worldwide; its maximum reproduction is in the winter season. Its fruits are adhesives and odder, and its essential oils are used as colorants. Among the most outstanding uses are the fodder resource and the medicinal anti-inflammatory effect, inhibition with an ethanolic extract of Vibrio cholera, and anti-ulcerative, among other effects. In addition, its fruits have been used as unconventional feeding strategies for goats to transfer phenolic compounds with antioxidant activity to improve the quality of animal products (milk and cheese). In 2020, supplementation in a murine model induced obesity, where the incorporation of goat milk evidenced an increase in energy expenditure and oxygen volume modifying the body composition of the mouse, compared to a high-fat diet, demonstrated a biotransfer of bioactive compounds from VF present in the milk to the mouse model. Previously, this research group had evaluated the antioxidant and anti-inflammatory power of various polyphenol extracts of this plant resource. Additionally, several phenolic compounds present in the leaves, stems, bark, flowers, roots, and fruits of VF have been described, such as gallic acid, quercetin, methyl gallate, myricetin, naringenin, ferulic acid, kaempferol, among others.

Among the unique polyphenols in VF fruits are gallic acid, quercetin, and epicatechin. Previous studies have described the effect of these compounds in inhibiting enzyme activity, which could be used as an alternative to control postprandial blood glucose levels and thus reduce the risk and incidence of DM2. In 1989 Wadood and collaborators tested the effect of Acacia seed powder supplementation using an animal model (rabbits), demonstrating that a dose of 2.3 and 4 g/kg significantly reduced blood glucose levels; in this trial, a stimulant of insulin secretion by the beta cells of the pancreas (sulfonylurea) was used as a positive control.

Ogawa and collaborators had recently conducted clinical trials, reporting in different scientific reports, where the effect of the consumption of a polyphenolic extract of A. meansi during an initial period of 4 to 8 weeks of administration; and later in a subsequent trial to extend the administration time up to 12 weeks; reporting an essential response on glycemia in patients with glucose intolerance, improving the oral glucose curve in 90 and 120 minutes, being much more relevant the results when the period of consumption of the extract was extended up to 12 weeks; where the levels of glucose in fasting decreased, concerning the control group, being this effect significant with the reduction of the stories of glycosylated hemoglobin; without the presence of any adverse effect. It is essential to point out that the first trial (with 4 to 8 weeks of intervention) used a concentration of 250 mg of polyphenolic extract per capsule and administered four capsules/day/person (1,000 mg/d). For the second intervention, the trial (12 weeks); being the concentration of polyphenols per capsule was very similar to the previous test (245 mg/capsule), but this time six capsules (1470 mg/d) per day were administered to each participant.

Research questions:

1. Will the dose of 1.2 mg/kg of the polyphenolic extract of Vachellia farnesiana reduce the mean value of the area under the glycemic response curve of healthy volunteer subjects concerning a control group?
2. Will the dose of 1.2 mg/kg of the polyphenolic extract of Vachellia farnesiana affect the mean values of serum liver enzymes and urine biomarker KIM-1 in healthy volunteer subjects relative to a control group?

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form
2. Characteristics of interest

   * Healthy volunteer subjects over 18 years of age and under 50 years of age
   * Men or women
   * Body mass index (BMI): greater than 18.5 and less than 24.9 kg/m2
   * Fasting glucose: 70-100 mg/dL
   * Alkaline phosphatase (ALP): 44 to 147 IU/L
   * Alanine aminotransferase (ALT): 5 to 77 IU/L
   * Aspartate aminotransferase (AST): 8 to 33 IU/L
   * Total bilirubin: 1.2 mg/dL
   * Indirect bilirubin: 0.2-0.7 mg/dL
   * Creatinine in blood: 0.06-1.3 mg/dL
   * Able to give written informed consent

Exclusion Criteria:

* Kidney disease diagnosed by a physician
* Diabetes Mellitus 2 diagnosed by a physician
* Ingestion of over-the-counter or prescription medications. Allopathic/ayurvedic/homeopathic/centrally acting appetite suppressants in recent months.
* Bariatric surgery (gastric bypass, sleeve gastrectomy, adjustable gastric banding, biliopancreatic diversion with duodenal switch, etc.)
* Subjects on an extreme diet or exercise regimen (>8 hours).
* Smokers (> two cigarettes per day)
* Patients with alcohol abuse (>3 glasses per day or >7 drinks per week).
* Subjects with HbA1c greater than 6.5%.
* Subjects with clinically diagnosed arterial hypertension (BP) and BP >140/90 mm Hg.
* Subjects with diseases of the thyroid gland.
* Weight loss greater than 5% during the last six months
* Pregnant/lactating women.
* Subjects who do not give their consent to participate in the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-04-06 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Safety of the experimental beverage intake in healthy adults | Baseline and post intake
  Safety was assessed through liver and kidney profiles (serum/urine) and adverse event questionnaires, with comparison to the control group.
Impact of the experimental beverage on glycemic response. | One time only by participant
  Changes in glucose and insulin concentration during the oral glucose tolerance test after consumption of the experimental beverage compared to the control group.

SECONDARY OUTCOMES:
Blood glucose fasting | Baseline and 72 hours post consumption of the experimental beverage.
  Change in glucose concentration (mg/dL)
Oral glucose tolerance test | One-time assessment at visit 2
  Changes in glucose concentration at 20, 40, 60, 90 and 120 minutes (mg/dL)
Changes in Incretin hormone | One-time assessment at visit 2
  Changes in concentration of the incretin hormone (GLP-1 active and GIP; pg/mL), were measured using a Milliplex metabolic assay.
Liver function test in serum | Baseline and 72 hours post consumption of the experimental beverage.
  Variations in liver function markers: Aspartate aminotransferase, alanine aminotransferase, phosphatase alkaline (UI/L), indirect bilirubin, direct bilirubin and total bilirubin (mg/dL) were measured with a Beckman Coulter automatized system.
Serum kidney function | Baseline and 72 hours post consumption of the experimental beverage.
  Changes in kidney function markers: creatinine (mg/dL) were measured with a Beckman Coulter automatized system.
Urine kidney biomarker | One-time assessment at visit 3
  Changes in the concentration of the biomarker KIM-1 (mg/min) were measured using ELISA Kit.
Serum total polyphenol and antioxidant activity | One-time assessment at visit 2
  Serum average concentration of total polyphenol (umol GAE/L) and antioxidant activity (DPPH and ORAC, TE mM)

IPD SHARING:
Plan to Share IPD: No
No, The IPD is not be shared with other researchers

REFERENCES:
- [Background] Delgadillo Puga C, Cuchillo-Hilario M, Navarro Ocana A, Medina-Campos ON, Nieto Camacho A, Ramirez Apan T, Lopez-Tecpoyotl ZG, Diaz Martinez M, Alvarez-Izazaga MA, Cruz Martinez YR, Sanchez-Quezada V, Gomez FE, Torre-Villalvazo I, Furuzawa Carballeda J, Camacho-Corona MR, Pedraza-Chaverri J. Phenolic Compounds in Organic and Aqueous Extracts from Acacia farnesiana Pods Analyzed by ULPS-ESI-Q-oa/TOF-MS. In Vitro Antioxidant Activity and Anti-Inflammatory Response in CD-1 Mice. Molecules. 2018 Sep 18;23(9):2386. doi: 10.3390/molecules23092386. PMID 30231503
- [Background] Hernandez-Garcia E, Garcia A, Avalos-Alanis FG, Rivas-Galindo VM, Delgadillo-Puga C, Camacho-Corona MDR. Nuclear magnetic resonance spectroscopy data of isolated compounds from Acacia farnesiana (L) Willd fruits and two esterified derivatives. Data Brief. 2018 Dec 7;22:255-268. doi: 10.1016/j.dib.2018.12.008. eCollection 2019 Feb. PMID 30591945
- [Background] Delgadillo-Puga C, Cuchillo-Hilario M, Leon-Ortiz L, Ramirez-Rodriguez A, Cabiddu A, Navarro-Ocana A, Morales-Romero AM, Medina-Campos ON, Pedraza-Chaverri J. Goats' Feeding Supplementation with Acacia farnesiana Pods and Their Relationship with Milk Composition: Fatty Acids, Polyphenols, and Antioxidant Activity. Animals (Basel). 2019 Aug 1;9(8):515. doi: 10.3390/ani9080515. PMID 31374913
- [Background] Hernandez-Garcia E, Garcia A, Garza-Gonzalez E, Avalos-Alanis FG, Rivas-Galindo VM, Rodriguez-Rodriguez J, Alcantar-Rosales VM, Delgadillo-Puga C, Del Rayo Camacho-Corona M. Chemical composition of Acacia farnesiana (L) wild fruits and its activity against Mycobacterium tuberculosis and dysentery bacteria. J Ethnopharmacol. 2019 Feb 10;230:74-80. doi: 10.1016/j.jep.2018.10.031. Epub 2018 Oct 25. PMID 30367988